CLINICAL TRIAL: NCT02035280
Title: Prospective Evaluation of Elderly Deformity Surgery: A Prospective Observational, Multicenter Study
Brief Title: Prospective Evaluation of Elderly Deformity Surgery
Status: Completed | Type: Observational
Sponsor: AO Foundation, AO Spine (Other)
Collaborators: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Other Study IDs: PEEDS
Record Dates: First submitted 2013-12-19; First posted 2014-01-14 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Adult Spinal Deformity
Keywords: Spine; Deformity; Fusion; Elderly; SRS-22r
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Elderly suffering of spine deformity: Spinal deformity patients over the age of 60 years undergoing elective surgery and requiring fusion of at least 5 levels.

SUMMARY:
As the population continues to age, the prevalence of spinal deformity surgery for older patients is increasing. Questions regarding the suitability of these patients to undergo large spinal procedures and whether the outcomes merit the risks involved are not well known.

DETAILED DESCRIPTION:
225 subjects greater than or equal 60 years of age with moderate and severe adult spinal deformity requiring surgical correction will be enrolled in a prospective multicenter international study. Spinal deformity will be defined as any coronal or sagittal plane spinal deformity in patients who have not undergone any previous spinal surgery (with the exception of prior decompression of a maximum of 2 levels) necessitating at a minimum a 5-level spinal fusion procedure. Standard radiographs and cross sectional imaging will be performed preoperatively, postoperatively, at 24 months and 5 years after surgery. Preoperative disease specific and general health questionnaires will be completed by all patients (EQ-5D, ODI, SRS-22r, NRS for back and leg pain). Follow up visits with questionnaires will be performed at 10 weeks (± 6 weeks), 12 months (± 2 months), 24 months (± 2 months) and 5 years (±6 months) post-operatively. All treatment-related AEs will be documented.

Regression analyses will be used to evaluate the association between patient demographics, comorbidities, treatment history, spinal deformity characteristics, surgical characteristics, treatment-related AEs and pre-surgical status to self-reported and radiographic outcomes after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older at the time of surgery
* Diagnosis of adult spinal deformity either in the coronal or sagittal plane requiring at the minimum a 5-level spinal fusion procedure
* Ability to understand the content of the patient information / Informed Consent Form
* Willingness and ability to participate in the clinical investigation according to the Clinical Investigation Plan (CIP)
* Signed and dated Institutional Review Board (IRB)/Ethics Committee (EC)-approved written informed consent
* Reconsent of patients for the 5 year follow-up if required by the IRB/EC

Exclusion Criteria:

* Any previous spinal procedure (except prior decompression of a maximum of 2 levels)
* Neurodegenerative disease or paralysis
* Unlikely to comply with follow-up
* Institutionalized individuals
* Any not medically managed severe systemic disease
* Recent history (≤ 3 months) of substance abuse (ie, recreational drugs, alcohol) or psychosocial disturbance that would preclude reliable assessment
* Prisoner
* Presence of active malignancy
* Has active, overt bacterial infection, systemic or local
* History of recent(≤ 3 months) fracture/malignancy in the spinal region
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly patients undergoing elective surgery for spinal deformity
Sampling Method: Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2013-12; Primary Completion 2021-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Absolute change in the Scoliosis Research Society-22 r (SRS-22r) total score | Baseline, 10 weeks, 12 months, 24 months
  The primary outcome is the absolute change in the SRS-22r total score between baseline and 24-months follow-up (FU) values in patients at age 60 or older treated with major spinal reconstruction.
  The SRS-22r is a patient-reported outcome instrument and has a range from 1 (worst) to 5 (best). It contains 22 questions covering five domains: function, pain, self-image, mental health (each with 5 items), and satisfaction with treatment (2 items) and each item is scored from 1 to 5.

SECONDARY OUTCOMES:
Treatment-related adverse events | Surgery, 10 weeks, 12 months, 24 months, 5 years
Oswestry Disability Index Version 2.1a (ODI) | Baseline, 10 weeks, 12 months, 24 months, 5 years
  The outcome measure is the absolute change between baseline, the 24-month and the 5-year FU values.
  The ODI is a patient-reported outcome measure used most commonly in patients with low back pain. It consists of 10 questions and each of the items can be scored from 0 (no disability) to 5 (maximal disability), leading to a maximum score of 50.
EuroQoL5 (EQ-5D). | Baseline, 10 weeks, 12 months, 24 months, 5 years
  The EQ-5D is a standardized instrument designed for self-completion to assess quality of life. It has 5 items with a three-point categorical response scale. A unique EQ-5D health state is defined by combining one level from each of the five dimensions.
  The EQ-5D is a standardized instrument designed for self-completion to assess quality of life. It has 5 items with a three-point categorical response scale. A unique EQ-5D health state is defined by combining one level from each of the five dimensions.
Pain (back and pain) | Baseline, 10 weeks, 12 months, 24 months, 5 years
  The outcome measure is the absolute change between baseline,the 24-month and 5 year FU values.
  Lower back and leg pain will be assessed on a visual analogue scale (NRS) which ranges from 0 (no pain) to 100 (severe pain).
Bone Mineral Density (BMD) | Baseline
  Baseline dual energy x-ray absorptiometry (DXA) scans of patients' BMD will only be performed at clinics where assessed as standard of care.
Radiological Parameters | Baseline, Surgery, 24 months, 5 years
  Radiological paramaters (lumbar lordosis, thoracic kyphosis, sagittal vertical axis, Cobb angle) will be measured at one pre- and two post-OP timepoints from sagittal standing and coronal standing x-rays.
Animal Fluency Test | Baseline, 10 weeks, 12 months, 24 months, 5 years
  The animal fluency test is a diagnostic tool that is recommended for use in clinical practice for quick assessment of cognitive impairment. The patient names as many animals as possible within a 60-second time period. Fifteen or fewer animals may indicate development of cognitive impairment.
SRS-22r | 5 years
  The SRS-22r is a patient-reported outcome instrument and has a range from 1 (worst) to 5 (best). It contains 22 questions covering five domains: function, pain, self-image, mental health (each with 5 items), and satisfaction with treatment (2 items) and each item is scored from 1 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lewis, MD, Principal Investigator — University of Toronto; Sigurd Berven, MD, Principal Investigator — University of California, San Francisco
Locations (13):
- United States (5):
  - UCSF Medical Center, San Francisco, California
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University Orthopedics, St Louis, Missouri
  - New York Presbyterian - Columbia University Medical Center, New York, New York
  - University of Virginia, Charlottesville, Virginia
- Toronto Western Hospital, Toronto, Ontario, Canada
- China (2):
  - Queen Mary Hospital, Hong Kong
  - Nanjing University Medical School, Nanjing
- Rigshospitalet, Copenhagen, Denmark
- Hamamatsu University School of Medicine, Hamamatsu, Japan
- St. Maartens Kliniek, Nijmegen, Netherlands
- Hospital Vall d'Hebron, Barcelona, Spain
- Aciboden Maser Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Campos Daziano M, Daunt L, Vashishth V, Seider E, Abbas A, Rienmueller A, Matsuyama Y, Qiu Y, Kelly M, Smith JS, Dahl BT, Spruit M, de Kleuver M, Polly DW, Sembrano J, Pellise-Urquiza F, Cheung KMC, Alanay A, Lenke LG, Shaffrey CI, Berven SH, Lewis SJ; PEEDS Study Group and AO Spine Knowledge Forum Deformity. Can Social Function Improve in Older Patients Undergoing Multi-Level Spinal Deformity Surgery? Global Spine J. 2025 Dec 27:21925682251411237. doi: 10.1177/21925682251411237. Online ahead of print. PMID 41454904